CLINICAL TRIAL: NCT06204029
Title: Everyone Can Sing. A Feasibility Study of Class Choir as a Mental Health Promoting Intervention Among 0-3rd Grade Students
Brief Title: Everyone Can Sing: A Feasibility Study of a Mental Health Promoting Intervention Among 0-3rd Grade Students
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Southern Denmark (Other)
Collaborators: TrygFonden, Denmark (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 23/24953
Record Dates: First submitted 2023-12-12; First posted 2024-01-12 (Actual); Last update posted 2024-12-18 (Actual); Status verified 2024-12

CONDITIONS: Mental Health
Keywords: Mental Health; Students; Teachers; Primary School; Mental health promotion; Intervention; Feasibility study; Denmark
MeSH Terms: conditions — Psychological Well-Being

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Everyone can sing (Experimental): Students from 0-3rd grade receive class choir two lessons every week as part of their regular school schedule
  Interventions: Behavioral: Everyone can sing

INTERVENTIONS:
Behavioral: Everyone can sing — The choir lessons are taught by a trained choir leader in close collaboration with the teacher in each class. The choir leaders and music teachers at the school also facilitate choir in the morning for selected or all classes. A special AKS pedagogy is developed and based on the inclusive nature of joyful musicking with body and voice. The pedagogy is developed to ensure that everyone is taken care of, so all children regardless of social or cultural background develop social and professional competencies central to a positive school life. The most important elements in this pedagogy include: A co-teacher system; Each student has a "choir partner"; Discipline in the classroom lessons is maintained by clear, simple, and subtle means.

SUMMARY:
This study aims to explore the feasibility of implementing and evaluating a class-based intervention in three Danish primary schools. The intervention includes class choir among all students in 0 to 3rd grade as part of the regular school schedule.

DETAILED DESCRIPTION:
Approximately every fifth child in Denmark experience mental health problems, mental illness, or low levels of school thriving before the age of ten, and 15% of Danish adolescent are diagnosed with a mental disorder before they turn 18. The experience of mental health problems, low school thriving and mental illness in childhood and adolescence is a severe risk factor for school segregation, low grades, school dropout and mental illness in youth and adulthood. There is therefore an urgent need for feasible and effective mental health promoting and preventive interventions from early childhood. High-quality music singing (e.g. choir singing) can promote well-being, social inclusion in school, and positive social relations among school-children, which are key prerequisites for strengthening children's mental health. However, the potential benefits of this type of intervention have not been evaluated in a Danish context. Therefore, we developed the Alle kan synge (AKS; in English: Everyone can sing) intervention as a prototype for implementation and dissemination.

The aim of this feasibility study is to explore the feasibility of implementing the AKS intervention in three Danish primary schools and assess feasibility of the evaluation design. Findings will provide knowledge on the critical aspects of the intervention, which may lead to a possible refinement of the AKS intervention, the implementation processes or evaluation design.

ELIGIBILITY:
Inclusion Criteria: All students in grades 0 to 3 (typically aged 5 to 10 years) in three different Danish elementary schools

Exclusion Criteria: None

Ages: 5 Years to 10 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 910 (Actual)
Dates: Start 2024-01-04 (Actual); Primary Completion 2025-03 (Estimated); Study Completion 2025-03 (Estimated)

PRIMARY OUTCOMES:
Mental Health. It will be completed by the student's parents and schoolteacher. | Measurements at baseline and 1-year follow-up
  Measured by the Strengths and Difficulties Questionnaire (SDQ). SDQ consists of 25-items rated on a 3-point Likert scale (not true, somewhat true, and certainly true), with a positive and negatively phrased items. 'Somewhat True' is always scored as 1, but the scoring of 'Not True' and 'Certainly True' varies with the item. The SDQ can be divided between five sub-scales (five questions each): Emotional Symptoms, Conduct Problems, Hyperactivity-Inattention, Peer Problems, Pro-Social Behaviour. Total Difficulties Score is adding scores from all scales except the prosocial scale (score range 0-40). Higher scores represent more problems. This is supplemented with a brief impact supplement, where items on distress and impairment can be added up to generate an impact score that ranges from 0 to 10 for parent-report, and from 0 to 6 for teacher-report.

SECONDARY OUTCOMES:
Mental health. It will be completed by the students. | Measurements at baseline and 1-year follow-up
  Measured with the five items of the World Health Organisation Five Well-Being Index (WHO-5). Response options range from 0 (Never) to 4 (All of the time): Total score range of 0-20 with higher values indicate higher mental well-being. In addition, one item about wellbeing: "That's how I feel most of the time" with responses from very happy to not happy and one item bout general self-efficacy: "Are you good at solving your problems".
School thriving. It will be completed by the students. | Measurements at baseline and 1-year follow-up
  Measured by one item regarding the general feeling about school and two indicators of not thriving: Do you have stomach aches at school? Do you have headaches at school? I
Class coherence. It will be completed by the students. | Measurements at baseline and 1-year follow-up
  Measured by four items regarding 1) I like my class, 2) students in the class are helpful, 3) students in the class enjoy being together, and 4) I believe the others in the class like me.
Social inclusion. It will be completed by the students. | Measurements at baseline and 1-year follow-up
  Assessed through four items: 1) Do you feel alone at school, 2) Do you get teased at school, so it makes you feel sad, 3) Who from the class do you play with the most during recess, 4) If you could decide for yourself: Who would you like to sit next to in class.

CONTACTS AND LOCATIONS:
Overall Officials: Katrine R Madsen, Principal Investigator — University of Southern Denmark
Locations (1):
- University of Southern Denmark, Copenhagen, Denmark

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Madsen KR, Tetens A, Bonde LO, Kusier AO, Jeppesen P, Andersen S. Everyone Can Sing: Protocol for a non-randomized feasibility study of class choir as mental health promotion among primary school children (ages 5-10) in Denmark. Pilot Feasibility Stud. 2025 Dec 31. doi: 10.1186/s40814-025-01757-8. Online ahead of print. PMID 41469714